CLINICAL TRIAL: NCT00000401
Title: Open Label Multicenter Induction of CII Tolerance in Patients With Rheumatoid Arthritis
Brief Title: Oral Collagen for Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Arnold E. Postlethwaite, MD, University of TN Health Science Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AR045255 (NIH); R01AR045255 (NIH); NIAMS-037
Expanded Access: Available
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Rheumatoid Arthritis
Keywords: NSAIDs; Oral Tolerance; Drug Interaction; Oral Administration; Interleukin 10; Collagen; Chemotherapy; Human Therapy Evaluation; DMARDs; RA; IL-10
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The low dose group will receive CII 30 mcg daily for 10 weeks, then 50 mcg daily for 10 weeks, followed by 70 mcg daily for 10 more weeks.
  Interventions: Drug: Oral bovine type II collagen
- 2 (Experimental): The high dose group will receive CII 90 mcg daily for 10 weeks, then 100 mcg daily for 10 weeks, followed by 130 mcg daily for 10 more weeks.
  Interventions: Drug: Oral bovine type II collagen

INTERVENTIONS:
Drug: Oral bovine type II collagen — Drug can be interrupted or stopped for suspected adverse events.
  Other Names: CII

SUMMARY:
Rheumatoid arthritis (RA) is an autoimmune disease characterized by swelling and inflammation of the joints. In RA, the immune system attacks a person's own cells inside joints, eventually leading to joint damage and disability. This study will determine if oral bovine type II collagen (bovine CII) will lead to decreased joint inflammation in RA patients.

DETAILED DESCRIPTION:
RA is an inflammatory disease that causes pain, swelling, stiffness, and loss of function in the joints. The study will evaluate the effects of using oral bovine CII on RA patients by assessing the levels of inflammation markers such as interferon gamma (IFN-gamma), interleukin-10 (IL-10), and transforming growth factor beta (TGF-beta). This study is a multicenter clinical trial to be conducted at the University of Tennessee, Memphis (the lead center) and the West Tennessee Medical Specialty Clinic (a collaborating site).

Patients enrolled will be allowed to continue a constant dose of disease-modifying anti-rheumatic drugs (DMARDs) and prednisone less than or equal to 7.5 mg/day. Patients will be randomly assigned to one of two groups. The low dose group will receive 30 mcg daily for 10 weeks, then 50 mcg daily for 10 weeks, followed by 70 mcg daily for 10 more weeks; the high dose group will receive 90 mcg daily for 10 weeks, then 100 mcg daily for 10 weeks, followed by 130 mcg daily for 10 more weeks. Blood will be collected at screening and at Weeks 10, 20, and 30. Blood will be analyzed for indicators of inflammation.

Note: this trial is no longer being conducted as an intervention trial. Accrual has been discontinued, although patients previously enrolled are still being followed.

ELIGIBILITY:
Note: accrual into this trial has been discontinued, but patients previously enrolled are still being followed.

Inclusion Criteria:

* Clinically stable RA and unlikely to require adjustment of doses of DMARDs, NSAIDs, prednisone, or anti-TNFα therapies for the treatment phase of the study
* Meets American College of Rheumatology (ACR) 1988 revised criteria for RA
* Onset of disease at age 16 or older
* Onset of disease at least 3 months prior to enrollment
* PBMC - IFNγ - α1(II)/PBS stimulation index greater than or equal to 1.5 in 6 months prior to baseline visit
* Agree to discontinue herbal remedies described in this protocol
* Agree to use acceptable forms of contraception

Exclusion Criteria:

* Participation in another clinical research study involving the evaluation of another investigational drug within 90 days prior to study entry
* Currently taking greater than 7.5 mg prednisone daily
* Intra-articular corticosteroid injections within 30 days prior to study entry
* Concurrent serious medical condition which, in the opinion of the investigator, makes the patient inappropriate for the study
* Pregnancy
* Beef allergy
* Use of fish oil within 4 weeks of study entry
* Previous use of auranofin or cyclophosphamide (all other DMARDs are allowed)
* Previous autologous or heterologous stem cell transplantation
* Active malignancy or past treatment consisting of antineoplastic drugs or total lymphoid irradiation
* Intolerance to citrus juices or colorless carbonated beverages

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 1999-07; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Repeated measures analysis of variance with contrasts to determine if the change in the PBMC-IFN gamma-alpha 1(II)/PBS stimulation index is significantly at the 0.05 level and/or greater than or equal to 30%. | Before and after each 10-week treatment

SECONDARY OUTCOMES:
A Pearson correlation coefficient will be calculated for the change in the PBMC-INF gamma-alpha1(II)/PBS stimulation index and the change in the reactivity to RA CII epitope alpha 1 (II) CB11 for each dose. | Before and after each 10-week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Arnold E. Postlethwaite, MD, Principal Investigator — University of Tennessee at Memphis Department of Medicine
Locations (2):
- United States (2):
  - The Arthritis Clinic of Jackson, PLLC, Jackson, Tennessee
  - University of Tennessee, Memphis, Memphis, Tennessee

REFERENCES:
- [Background] Postlethwaite AE. Can we induce tolerance in rheumatoid arthritis? Curr Rheumatol Rep. 2001 Feb;3(1):64-9. doi: 10.1007/s11926-001-0052-z. PMID 11177772
- [Result] Carbone LD, McKown K, Pugazhenthi M, Barrow KD, Warrington K, Somes G, Postlethwaite AE. Dosage effects of orally administered bovine type I collagen on immune function in patients with systemic sclerosis. Arthritis Rheum. 2004 Aug;50(8):2713-5. doi: 10.1002/art.20361. No abstract available. PMID 15334493